CLINICAL TRIAL: NCT04018157
Title: Single Bolus Dose of Ketodex Versus Ketofol For Prevention Of Emergence Agitation In Adults Undergoing Nasal Surgeries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, olfat abd elmoniem ibrahem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5452
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Agitation, Emergence
Keywords: ketodex, ketofol , agitation , nasal surgery
MeSH Terms: conditions — Emergence Delirium; Psychomotor Agitation | interventions — Ketamine; Dexmedetomidine; Propofol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: patient and outcomes assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ketodex (Active Comparator): ketamine dexmedetomidine mixture
  Interventions: Drug: "Ketamine" and "dexmedetomidine" and "propofol" and "0.9%saline"
- ketofol (Active Comparator): ketamine propofol mixture
  Interventions: Drug: "Ketamine" and "dexmedetomidine" and "propofol" and "0.9%saline"
- placebo (Placebo Comparator): normal saline
  Interventions: Drug: "Ketamine" and "dexmedetomidine" and "propofol" and "0.9%saline"

INTERVENTIONS:
Drug: "Ketamine" and "dexmedetomidine" and "propofol" and "0.9%saline" — patients will receive single intravenous bolus of combination from ketamine 0.5mg/kg and dexmedetomidine 1ug/kg in one syringe diluted in 10 ml 0.9% saline.
  Other Names: ketalar; precedex; diprivan

SUMMARY:
* emergence agitation is seen in around 68% after nasal surgeries. Agitated patients needs more staff and nurses to control their abnormal movement which leads to self extubation , removal of catheters and bruises in the extremities.
* Dexmedetomidine, ketamine, propofol intravenous infusion and other agents was used to prevent EA . Recently, ketodex is found to reduce the incidence and severity of EA .
* We aim to compare single bolus dose of Ketodex Versus Ketofol For Prevention Of emergence Agitation in adults undergoing nasal surgeries.

DETAILED DESCRIPTION:
The incidence of emergence agitation (EA) after nasal surgeries is relatively high , it is reported to be 68% (1).The precise mechanism is not known. Awake extubation after nasal surgeries is preferred as the airway may be contaminated by blood , and the nasal airway may be blocked by surgical packs that causes sense of suffocation. Awake extubation and nasal pack is a trigger to emergence agitation(2).

emergence agitation (EA) is harmful to the patient and the staff, it Characterized by disorientation, confusion, abnormal violent movement that may result in serious complication and morbidity(3). It develops early with the recovery from general anesthesia(4). Although agitation is more observed in pediatrics but its incidence in adults reach up to 21.4% (5).

Different medication agents such as anesthetic drugs, benzodiazepine and α2 agonist was proved to attenuate the EA with different efficiencies (6).

Dexmedetomidine is a selective α2 adrenoceptor agonist. It has sedative, hypnotic, anxiolytic, analgesic and sympatholytic properties. It was proved to reduce the EA in children(7). However there was few data about its effect in reducing the agitation in adult after general anesthesia(8).

Propofol is short acting hypnotic and sedative agent. It is used for induction and maintenance of anesthesia(9). Previous studies proved that propofol was effective in preventing EA (10,11) and depends on the time of administration(12).

Ketamine is N-methyl- D-asparate receptor antagonist, it has anesthetic, sedative and analgesic effect(13).

Ketofol is a combination of low dose ketamine with propofol , it has been used for sedation and analgesia. The effect of this combination was supposed to produce less toxicity compared to each drug alone by decreasing the required doses(14).

Ketodex is combined low dose of ketamine and dexmedetomidine, it was used for sedation , this combination decrease some of the pitfalls occurring when use dexmedetomidine as a sole agent(15).

Most EA studies was done in pediatric. To our knowledge there was no previous studies report the effect of bolus dose of ketodex versus ketofol on the incidence and prevention of EA after nasal surgeries in adults. This study aimed to compare single bolus dose of Ketodex Versus Ketofol For Prevention Of Emergence Agitation In adults Undergoing nasal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.

  * Both gender.
  * Age (21-60) years old.
  * patient with Body Mass Index (BMI) (25-35kg/m²).
  * American Society of Anesthesiologist (ASA) I / II
  * Adult patient scheduled to elective nasal surgeries

Exclusion Criteria:

* - Patient with difficult airway (mallampati III,IV).
* Altered mental status (psychiatric and anxiety disorder).
* Post traumatic stress disorders.
* History of allergy to study drugs.
* Patient on sedative or hypnotic medication.
* Patients with chronic pain or on painkiller.
* Patients with severe hepatic or kidney impairment.
* Patients having a history of thyrotoxicosis, hypertension, cardiac , chest or neurological disease.
* Patient receiving B agonist.
* Pregnant or breast feeding female.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-23 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence agitation. | up to 60 minutes after extubation
  The incidence of emergence agitation.
The level of emergence agitation. | up to 60 minutes after extubation
  The level of emergence agitation measured by . Richmond Agitation-Sedation scale (RASS) is ten scales; five for sedation level ,one for alertness and calmness, and four for agitation level as follow: -5 unarousable , -4 deep sedation , -3 moderate sedation , -2 light sedation , -1 drowsy ; 0 alert and calm,+1 restless , +2 agitated , +3 very agitated and +4 combative. Patients with score ≥ 2 considered having agitation.

SECONDARY OUTCOMES:
The Emergence time | up to 20 minutes after discontinuation of isoflurane
  The time from discontinuation of isoflurane to first response to verbal command.
The extubation time | up to 20 minutes after discontinuation of isoflurane
  time from discontinuation of isoflurane to extubation.
The time of discharge | up to 40 minutes after extubation
  The time from arrival to postanesthesia care unite (PACU) to discharge to the ward according to modified aldert score
Postoperative Pain is evaluated using Numerical rating Scale (NRS) | up to 40 minutes after extubation
  (NRS) A commonly used scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border.
"Number of Participants with vomiting or hypotension or bradycardia" | all over 40 minutes post-operative
  vomiting , hypotension, bradycardia Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Olfat Amin, M.D, Principal Investigator — Faculty of medicine, Zagazig university
Locations (1):
- Faculty of Medicine, Zagazig, Elsharkia, Egypt

IPD SHARING:
Plan to Share IPD: No